CLINICAL TRIAL: NCT01462058
Title: The Role of Vitamin D Supplementation on Well Being and Symptoms of Depression During the Winter Season in Health Service Staff
Acronym: D3-vit-SAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Connie Thuree Nielsen, consultant, MD, ph.d (Other)
Responsible Party: Sponsor-Investigator, Connie Thuree Nielsen, consultant, MD, ph.d, MD, ph.d, Region Syddanmark
Organization: Region Syddanmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ID-301115
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Seasonal Affective Disorder; Vitamin D3; Mental Health; Dietary Supplement
Keywords: SPAQ; Sigh-SAD; Hamilton 29; Vitamin D3; p25(OH)D
MeSH Terms: conditions — Seasonal Affective Disorder; Psychological Well-Being | interventions — Cholecalciferol; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Active Comparator): one tablet of vitamin D3 (70µg) per day for 12 weeks.
  Interventions: Dietary Supplement: Vitamin D3
- placebo (Placebo Comparator): one tablet of sugar pill per day for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 70µg Vitamin D3, daily, 12 weeks
  Other Names: Active
  Arms: Vitamin D3
Drug: Placebo — Placebo, daily, 12 weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to investigate whether vitamin D3 (70 micrograms) is better than placebo in preventing depression symptoms among employees in health care

DETAILED DESCRIPTION:
Vitamin D3 is produced in the skin after exposure to ultraviolet B light from the sun. Vitamin D3 is metabolised sequential in the liver into 25-hydroxy-vitamin D [25(OH)D], which is the storage form of vitamin D in the body, and then in the kidney into the steroid hormone, 1a,25-dihydroxyvitamin 1a,25-dihydroxyvitamin D [1,25(OH)2D].

At higher latitudes ultraviolet B light is stopped by the atmosphere during winter season. Half of Danes have low levels of [25(OH)D] in the blood and especially in the early spring months the levels of [25(OH)D] are low. In addition, Vitamin D3 is absorbed through the gut from vitamin D-rich food sources. But several studies show that it is not possible through a recommended diet, which consists of 300 g of fish per week to consume adequate amounts of vitamin D3.

New research suggests link between vitamin D3 and brain function.In the Central Nervous System (CNS) there are specific nuclear receptors for 1,25(OH)2D (VDR) and the enzymes necessary for the hydroxylation of 25(OH)D to 1,25(OH)2D are also present in CNS.

In clinical studies, low serum levels of 25(OH)D, have been associated with reduced cognitive function, anxiety and depression.

The objective of this randomized clinical trial is to investigate whether indoor employees, with tendency to depressive symptoms in the winter season, should be offered vitamin D3 supplements during the Winter season, or it has no significance in relation prevent depressive symptoms.

The study is carried out in the winter season in the Region of Southern Denmark for 12 weeks and offered to health service staff, who have a tendency for depressive symptoms in the winter season.

ELIGIBILITY:
Inclusion Criteria:

* Health service staff and employee in the Region of Southern Denmark.
* Tendency to depressive symptoms in the winter season SPAQ>7.

Exclusion Criteria:

* clinical diagnosis sarcoidoses
* tuberculosis
* bipolar affective disorder
* schizophrenia
* hypercalcemia
* hyperphosphatemia
* pregnancy
* hyperparathyroidism
* reduced kidney function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Hamilton-29 | 12 weeks
  Change from baseline in Hamilton-29 at week 12

SECONDARY OUTCOMES:
WHO-5 | 12 weeks
  Change from baseline in WHO-5 at week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Services Esbjerg, Esbjerg, Esbjerg N, Denmark

REFERENCES:
- [Derived] Frandsen TB, Pareek M, Hansen JP, Nielsen CT. Vitamin D supplementation for treatment of seasonal affective symptoms in healthcare professionals: a double-blind randomised placebo-controlled trial. BMC Res Notes. 2014 Aug 14;7:528. doi: 10.1186/1756-0500-7-528. PMID 25125215